CLINICAL TRIAL: NCT05029297
Title: Study of Efficacy and Non-inferiority, With Two Capsaicin Topic Treatments, for the Moderate to Severe Pain in Diabetic Neuropathy.
Brief Title: Study With Two Capsaicin Topic Treatments in Diabetic Neuropathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arafarma Group, S.A. (Industry)
Collaborators: Fundación Teófilo Hernando, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ITHUEC-CAP/10-5
Record Dates: First submitted 2021-05-19; First posted 2021-08-31 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Patients will receive one of the two interventions (CAPSAICIN topical solution and cream) during the initial phase of the study of 8 weeks and receive the other intervention during the second phase of the study of 8 weeks. Both phases will be separated in a 4 week washout period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPSAICIN 0.75 mg/g topical solution applicable in roll-on (Experimental): CAPSAICIN 0.75 mg / g topical solution applicable in roll-on: 4 applications per day for 8 weeks.
  Interventions: Drug: Capsaicin
- CAPSAICIN 0.075% cream (Active Comparator): CAPSAICIN 0.075% cream (ARAFARMADOL® 0.075% cream): 4 applications per day for 8 weeks.
  Interventions: Drug: Capsaicin

INTERVENTIONS:
Drug: Capsaicin

SUMMARY:
Clinical trial of "line extension" of drug ARAFARMADOL® 0.075% cream in a new formulation in topical solution applicable in roll-on and with the same therapeutic indications approved for the cream.

DETAILED DESCRIPTION:
The sponsor created a new pharmaceutical formulation of CAPSAICIN topical solution applicable in roll-on. This new formulation in roll-on represents a line extension of drug ARAFARMADOL 0.075 cream, which is currently marketed in Spain by the sponsor.

The proposed investigational product as topical solution applicable in roll-on is expected to solve the compliance and safety issues of the cream with the same indications for use.

Eligible patients will be randomized into two groups: CAPSAICIN topical solution applicable in roll-on and CAPSAICIN cream (ARAFARMADOL® ) for 8 weeks. Then, they will have a 4 week washout period and will be crossed over to the other treatment group for 8 weeks. A follow-up period of 2 weeks will take place after the end of both treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Written or oral informed consent with witnesses, before initiating the specific procedures of the protocol.
2. Non-pregnant, non-lactating man or woman ≥ 18 years.
3. Patients diagnosed with Type I or II Diabetes Mellitus, treated or untreated.
4. Patients with a diagnosis of painful peripheral diabetic neuropathy, treated or not treated
5. Painful diabetic neuropathy of at least 3 months of evolution with moderate to severe pain ≥ 4 on the VAS scale in the selection phase.
6. The pain must have been experienced daily, interfered with daily activities or sleep, and not attributable to psychological origin.
7. Stabilization of pain medication at least during the month prior to the start of treatment. The patient must be prepared to remain in treatment with the same pain medications at the same doses as previous to the start, during the study and in the follow-up phase (24 weeks).
8. Intact, non-irritated and dry skin in the painful areas to be treated.
9. Patients with the ability to collaborate in the trial.

Exclusion Criteria:

1. Allergic reactions to capsaicin.
2. Patients with neuropathic pain of an etiology other than diabetes.
3. Patients with peripheral ischemic pain due to diabetic artery disease.
4. Patients with unstable glycemic control (glycosylated Hb ≥ 10.5%).
5. Amputation of any part of the lower limb.
6. Surgery scheduled during the clinical trial.
7. Mild painful diabetic neuropathy (<4 VAS).
8. Other serious pathologies:

   * Documented congestive heart failure or systolic dysfunction (LVEF ≤ 50%).
   * Previous history of myocardial infarction in the 6 months prior to enrollment.
   * Uncontrolled hypertension (160/110 mmHg maximum).
   * Uncontrolled high-risk arrhythmias.
   * Significant neurological or psychiatric disorders, including psychotic disorders, dementia that prevent patients from understanding and giving informed consent.
   * Active uncontrolled infection.
9. Use other topical pain medications in painful areas.
10. History or current problem of substance abuse.
11. Pregnant or lactating women. Women of childbearing potential should use effective contraception.
12. Participation in another clinical trial with any non-marketed investigational drug during the 90 days prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-11-04 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy and the non-inferiority of a new formulation of the capsaicin topical solution in "roll-on" compared to capsaicin in cream. | Baseline to 8 weeks
  To demonstrate the efficacy and the non-inferiority of a new formulation of Capsaicin 0.75 mg / g topical solution applicable in "roll-on" compared to the formulation currently marketed (comparator) in cream (Arafarmadol® 0.075% cream). The main variable will be the decrease in pain on the visual analogue pain scale (score range from 0 (no pain) to 10 (worst pain possible) at 8 weeks of treatment with each drug. The change in efficacy between the two treatments (pain reduction with cream minus pain reduction with roll-on) will be calculated and the 95% confidence interval for this change will be obtained; If the confidence interval does not exceed the non-inferiority limit (1.0), it will be concluded that the new formulation is not inferior to the one currently marketed.

SECONDARY OUTCOMES:
Rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) between both treatment groups. | From Visit 1, and at each visit, up to 22 weeks.
  All AEs will be recorded, whether considered minor or serious, drug-related or not.
Change from baseline in both treatment groups of QoL. | Baseline to 8 weeks
  The EQ-5D consists of 2 parts - the descriptive part and the visual scale analog (EVA). The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, habitual activities, pain / discomfort, and anxiety / depression. In the EVA the patient scores their health between two extremes, 0 and 100, worst and best health status imaginable.
Treatment compliance in both treatment groups. | At the end of each treatment phase (8th week).
  Treatment compliance is measured by the use of Morisky-Green test.
Change from baseline in both treatment groups of height. | Baseline to every 4 weeks up to 22 weeks.
  Height measured by cm.
Change from baseline in both treatment groups of weight. | Baseline to every 4 weeks up to 22 weeks.
  Weight measured by kg.
Change from baseline in both treatment groups of blood pressure. | Baseline to every 4 weeks up to 22 weeks.
  Blood pressure measured by mm Hg.
Change from baseline in both treatment groups of dermatological assessment of the painful area. | Baseline to 8 weeks.
  Dermatological assessment is measured by Dermatological Assessment Scale (scale range from 0 (without causing irritation) to 7 (important reaction that extends beyond the assessed area).
Grade of compliance/complacency of treatment. | Last Follow-Up visit of the study (22nd week).
  A patient compliance questionnaire (6 questions) will be self-administered to the patient and must be completed during the follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Raffaelle Carraro, Principal Investigator — Hospital Universitario La Princesa. Madrid. Investigator Site Coordinator.

IPD SHARING:
Plan to Share IPD: No